CLINICAL TRIAL: NCT07235345
Title: To Investigate the Effect of Pulmonary Surfactant With Different Inspired Oxygen Concentrations on the Clinical Outcomes of Very Preterm Infants Under Non-invasive Assisted Ventilation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Falin (Other)
Collaborators: Zhumadian Central Hospital (Other); Zhengzhou Central Hospital (Other); Xinyang Central Hospital (Other); Xinxiang Central Hospital (Other); Nanyang Central Hospital (Other); Zhoukou Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Xu Falin, Chief Physician, Third Affiliated Hospital of Zhengzhou University
Organization: Third Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-242-01
Record Dates: First submitted 2025-09-21; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Neonatal Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High fraction of inspired oxygen (No Intervention): Parameters such as pressure and respiratory rate were set according to relevant clinical guidelines or expert consensus. The initial FiO2 was 21% when PEEP was ≥6 cmH2O, and FiO2 was adjusted according to the respiration and percutaneous oxygen saturation (SpO2) of the children to maintain SpO2 90%-94%. When FiO2 reached 30%, PS treatment was given (the initial dose was 200mg/kg, and the second or third dose of 100mg/kg could be repeated if necessary if the disease progressed). PS treatment should be given as early as possible within 6 hours after birth. Endotracheal intubation, INSURE technique, or LISA technique can be used.
- Low fraction of inspired oxygen (Experimental): Parameters such as pressure and respiratory rate were set according to relevant clinical guidelines or expert consensus. The initial FiO2 was 21% when PEEP was ≥6 cmH2O, and FiO2 was adjusted according to the respiration and percutaneous oxygen saturation (SpO2) of the children to maintain SpO2 90%-94%. PS was given when FiO2 reached 25% (the initial dose was 200mg/kg, and the second or third dose of 100mg/kg could be given if necessary if the disease progressed), and PS was administered as early as possible within 6 hours after birth. Endotracheal intubation, INSURE technique, or LISA technique can be used.
  Interventions: Other: According to the FiO2 threshold of PS application corresponding to randomization, PS treatment was given when FiO2 reached the threshold

INTERVENTIONS:
Other: According to the FiO2 threshold of PS application corresponding to randomization, PS treatment was given when FiO2 reached the threshold — According to the relevant clinical guidelines or expert consensus, the pressure, respiratory rate and other parameters were set. The initial FiO2 was 21% when PEEP was ≥6 cmH2O. FiO2 was adjusted according to the respiration and percutaneous oxygen saturation (SpO2) of the children. To maintain SpO2 90%-94%. According to the FiO2 threshold corresponding to randomization, PS treatment was given when FiO2 reached the threshold (the initial dose was 200mg/kg, and the second or third dose of 100mg/kg could be repeated if necessary if the disease progressed). PS treatment was administered as early as possible within 6 hours after birth. Endotracheal intubation, INSURE technique, or LISA technique can be used.
  Arms: Low fraction of inspired oxygen

SUMMARY:
A prospective multicenter randomized controlled study was conducted. Eligible very preterm infants with a gestational age of <32 weeks were enrolled. All infants received routine treatment after birth and were randomly divided into two groups according to the FiO2 threshold of PS under noninvasive assisted ventilation: Control group (FiO2=0.30) and low concentration group (FiO2=0.25). Clinical data were collected to explore the differences in clinical outcomes between the two groups.

DETAILED DESCRIPTION:
① All the very/extremely preterm infants who met the criteria were divided into low concentration group and high concentration group according to the random number table method. The pressure, respiratory rate and other parameters were set according to the relevant clinical guidelines or expert consensus. The initial FiO2 was 21% when PEEP was ≥6 cmH2O. To maintain SpO2 90%-94%. According to the FiO2 threshold corresponding to randomization, PS treatment was given when FiO2 reached the threshold (the initial dose was 200mg/kg, and the second or third dose of 100mg/kg could be repeated if necessary if the disease progressed). PS treatment was administered as early as possible within 6 hours after birth. Endotracheal intubation, INSURE technique, or LISA technique can be used.

② The basic information and perinatal outcomes of the two groups were collected; Outcome indicators: the main outcome indicators were the failure rate of non-invasive treatment, the time of tracheal intubation mechanical ventilation, the time of non-invasive assisted ventilation, the days of oxygen therapy, the time of the first use of PS, and the rate of repeated PS. The secondary outcomes included mortality, incidence of BPD, incidence of ROP, oxygen demand at 28 days after birth and 36 weeks of corrected gestational age, oxygen demand at discharge, length of hospital stay, and cost of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Very preterm infants with gestational age <32 weeks
* immediately transferred to the neonatal intensive care unit
* signs of respiratory distress or RDS requiring respiratory support;
* Informed consent was obtained from the families of the children.

Exclusion Criteria:

* Giving up treatment or being transferred to other hospitals during hospitalization;
* requiring mechanical ventilation with tracheal intubation immediately or within 2 hours after birth
* complicated with pneumothorax, complex congenital heart disease, congenital malformation, congenital cystic lung disease, chromosomal inherited metabolic diseases, etc
* Incomplete clinical data

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of tracheal intubation and mechanical ventilation | The children required tracheal intubation and mechanical ventilation during hospitalization, and the observation time was about 2 months
  The duration of invasive mechanical ventilation was observed
Time of first PS use | Time to first use of pulmonary surfactant within 6 hours after birth
  The time from the first use of PS to birth was observed
Duration of noninvasive assisted ventilation | Noninvasive ventilation was required during hospitalization, and the observation time was about 2 months
  The duration of noninvasive mechanical ventilation was observed during hospitalization
Repeat PS usage rate | The frequency of repeated use of pulmonary surfactant during hospitalization was observed for about 1 week after birth
  Whether PS was used repeatedly during hospitalization was observed
Days of Oxygen therapy | The children needed oxygen inhalation for a number of days during hospitalization, and the observation time was about 2 months
  The time of oxygen therapy during hospitalization was observed
Failure rate of noninvasive treatment | 72 hours after birth
  The use of invasive mechanical ventilation after birth was observed

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhengzhou University, Henan, Zhengzhou, China